CLINICAL TRIAL: NCT01164917
Title: A Randomized, Double-blind, Placebo-controlled, Single Dose, Two-period, Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Efficacy of AMG 811 in Subjects With Discoid Lupus Erythematosus
Brief Title: Safety Study of AMG 811 in Subjects With Discoid Lupus Erythematosus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The 16 subjects enrolled in the study should enable Amgen to adequately assess safety and tolerabili
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20100011
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Cutaneous Lupus; Discoid Lupus; Lupus; Systemic Lupus Erythematosus
Keywords: Lupus; Discoid Lupus; Cutaneous Lupus
MeSH Terms: conditions — Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AMG811 (Active Comparator): All will receive AMG 811, either on Day 1 or Day 85
  Interventions: Drug: AMG811
- AMG811 Placebo (Placebo Comparator): All will receive placebo, either on Day 1 or Day 85
  Interventions: Drug: AMG811 Placebo

INTERVENTIONS:
Drug: AMG811 — Twelve subjects will be randomized to receive AMG 811 in Period 1 and will receive AMG 811 Placebo in Period 2. The AMG 811 and AMG 811 Placebo will be administered by injection.
  Arms: AMG811
Drug: AMG811 Placebo — 8 subjects will be randomized to receive AMG 811 Placebo in Period 1 and will receive AMG 811 in Period 2. The AMG 811 Placebo and AMG 811 will be administered by injection
  Arms: AMG811 Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, two-period, crossover study in which approximately 20 subjects with Discoid Lupus Erythematosus will be enrolled to receive AMG 811 and placebo in one of two sequences (ie, AMG 811 followed by placebo or placebo followed by AMG 811).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between the ages of 18 and 70 years of age, inclusive, at the time of randomization;
* Diagnosis of discoid lupus erythematosus (DLE) with or without SLE;
* Intolerance of anti-malarial therapy or ≥ 3 months of anti-malarial therapy with residual disease activity. The total CLASI activity must be ≥ 10;
* Stable dose of topical steroids no stronger than medium-potency (Class III or less) for ≥ 2 weeks and/or systemic immunosuppressive therapy at stable dose for ≥ 8 weeks prior to randomization (except for leflunomide which requires ≥ 12 weeks) are permitted;
* Oral prednisone ≤ 20 mg/day (or equivalent) is permitted; one increase or one decrease of ≤ 5 mg/day prednisone equivalent (not to exceed 20 mg/day) will be allowed within 30 days before randomization;

Exclusion Criteria:

* Any disorder (including psychiatric), condition or clinically significant disease (other than a diagnosis of DLE or SLE) that would, by its progressive nature and/or severity, interfere with the study evaluation, completion and/or procedures per the investigator's discretion;
* History of malignancy;
* Signs or symptoms or relevant history of a viral, bacterial, fungal, and parasitic infection, or recent history of repeated infections;
* Subjects with evidence of past or active tuberculosis
* Positive serology for HIV antibodies, hepatitis B surface antigen or hepatitis C antibodies (confirmed by PCR or RIBA) during the screening period;
* Receipt of a live vaccine within 3 months of study randomization and during the study;
* Prior use of the following agents:
* Administration of an investigational biologic agent that primarily targets the immune system -
* Rituximab, Lymphostat-B, or TACl-Ig within 9 months prior to randomization (or comparable B cell depleting or B cell inhibiting biologics); Rituximab (or other depleting CD20 targeted agents) treated patients must demonstrate a return of CD19+ B cells to > 5/μL;
* CTLA4-Ig within 3 months prior to randomization;
* Other agents within 5 half-lives prior to randomization;
* Administration of cyclosporine, tacrolimus, sirolimus, IV immunoglobulin, and/or plasmapheresis within 3 months of randomization;
* Administration of thalidomide or lenalidomide within 3 months of randomization;
* Administration of oral or IV cyclophosphamide (or any other alkylating agent) within 9 months of randomization;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety evaluation: Subject incidence of treatment-emergent adverse events, clinically significant changes in vital signs, physical examination endpoints, clinical laboratory safety tests, ECGs and the development of anti-AMG811 antibodies | 197 days

SECONDARY OUTCOMES:
PK parameters, Change in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) score and IFN-gamma related gene expression in skin biopsy samples | 197 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (8):
  - Research Site, Santa Monica, California
  - Research Site, Stanford, California
  - Research Site, Atlanta, Georgia
  - Research Site, Ann Arbor, Michigan
  - Research Site, Durham, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Werth VP, Fiorentino D, Sullivan BA, Boedigheimer MJ, Chiu K, Wang C, Arnold GE, Damore MA, Bigler J, Welcher AA, Russell CB, Martin DA, Chung JB. Brief Report: Pharmacodynamics, Safety, and Clinical Efficacy of AMG 811, a Human Anti-Interferon-gamma Antibody, in Patients With Discoid Lupus Erythematosus. Arthritis Rheumatol. 2017 May;69(5):1028-1034. doi: 10.1002/art.40052. Epub 2017 Mar 31. PMID 28118537
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com